CLINICAL TRIAL: NCT05901337
Title: Influence of Cupping Therapy on Immune System in Post Covid- 19 Patients
Brief Title: Cupping Therapy on Immune System in Post Covid -19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Abd ElZahr, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: No:P.T.REC/012/003554
Record Dates: First submitted 2023-06-11; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Covid-19 Patients
MeSH Terms: interventions — Cupping Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cupping therapy with Convential medical treatment (Active Comparator): Cupping therapy with Convential medical treatment
  Interventions: Combination Product: Cupping therapy with convential medical treatment; Drug: Convential medical treatment
- Convential medical treatment (Active Comparator): Convential medical treatment
  Interventions: Combination Product: Cupping therapy with convential medical treatment; Drug: Convential medical treatment

INTERVENTIONS:
Combination Product: Cupping therapy with convential medical treatment — Device:Cupping therapy device
  Group A participants received Dry cupping therapy one session per week for 8 weeks with 6 days intervals between sessions and with cups applied to the skin for around 8 minutes. (In addition to convential medical treatment for 8 weeks in the form of :
  1. Vitamin D: The recommended dietary dose of vitamin D is 600 IU each day for adults 70 and younger .
  2. Vitamine C: The recommended dietary dose 200 mg/day vitamin c
  3. Anticoagulation drugs ("blood thinners")Doctors usually prescribe low-molecular-weight heparin (enoxaparin) (30 mg), each given subcutaneously every 12 hours .
Drug: Convential medical treatment — Group B participants received convential medical treatment for 8 weeks in the form of :
  1. Vitamin D: The recommended dietary dose of vitamin D is 600 IU each day for adults 70 and younger .
  2. Vitamine C: The recommended dietary dose 200 mg/day vitamin C
  3. Anticoagulation drugs ("blood thinners")Doctors usually prescribe low-molecular-weight heparin (enoxaparin) (30 mg), each given subcutaneously every 12 hours .

SUMMARY:
Purpose of this study is to investigate

1. The effect of Dry cupping therapy on T-Lymphocyte in post covid-19 patients.
2. The effect of Dry cupping therapy on serum Cytokine in post covid-19 patients.
3. The effect of Dry cupping therapy on Immunoglobulin IgA.
4. The effect of Dry cupping therapy on Immunoglobulin IgM.
5. The effect of Dry cupping therapy on Immunoglobulin IgG. seventy six patients of both genders with deficiency in T-Lymphocyte number,,higher level of serum cytokine and lower immunoglobulin IgA,IgM,IgG after two weeks of recovery from covid-19 . Age range from Twenty one to Sixty six years old .They participated in the study and recruited from surveillance unit of Shobra general hospital .These patients recruited by phone and have been offered to participate in the programme.The patients were divided equally into two groups (A and B). Assessment was done before and after treatment. T-Lymphocyte, serum cytokine and immunoglobulin IgA, IgM and IgG were analyzed by kenza 240 TX from fluorescence-labeled flow cytometry. Disposable cupping therapy instrument was used in treatment of group (A) in addition to traditional medical treatment in the form of vitamin C, D and anticoagulant drugs. Traditional medical treatment only was used in treatment of group (B).The obtained results of this study will determine the significant improvement of participated two groups.

   .

DETAILED DESCRIPTION:
Patient were selected randomly and distributed in two groups by computer generation. The sample size was calculated using the G*Power software (version 3.0.10). F-test MANOVA within and between interaction effects was selected. Considering a power of 0.80, an α level of 0.05 (2 tailed) and effect size of 0.39; two groups and response variables of five, a generated sample size of at least 38 participants per group was required and total sample size of 76 subjects.

ELIGIBILITY:
Inclusion Criteria:

* All patients with body mass index(BMI) 25.0-29.9 kg/m2 recruited two weeks post recovary from covid-19 and have lower T-lymphocyte and elevated cytokine All patients were clinically and medically stable.All patients recruited by phone and have been offered to participate in the programme.All patients will sign the informed consent before joining the study. Age range from 21 to 66 years .Subjects will be divided equally into two groups A,B. Assessment will be done before and after treatment.

Exclusion Criteria:

Patients will be excluded if they have any of the following criteria:

1. History of acute or chronic infections
2. Hepatobiliary diseases
3. Hematological diseases
4. Urinary system diseases
5. Nutrition and metabolism diseases
6. Rheumatic diseases
7. Endocrine diseases
8. Circulatory system diseases
9. Muscle trauma
10. Hypertension Further, if they fulfilled any of the following testing criteria
11. Hepatitis C virus antibodies
12. Human immunodeficiency virus antibodies
13. Creatinine above 120 μmol/L
14. Creatine kinase above 500 U/L
15. Uric acid above 475 μmol/L, glucose above 7.0 mmol/L
16. C-reactive protein above 12.0 m.

Ages: 21 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
T-lymphocyte | 3months
  1- Lymphocyte subset were analyzed from fluorescence-labeled flow cytometry on a DxFLEX flow cytometry by Kenza 240 Tx
Serum Cytokine | 3months
  Cytokine detection Kenza reagents were provided from a 240 TX bio lap diagnostic apparatus by microsphere flow immunofluorescence
ImmunoglobulinA,M,G | 3 months
  Kenza 240 TX for detection of immunoglobulin

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Mohamed, master, Principal Investigator — Physiotherapist at Shoubra general hospital
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No